CLINICAL TRIAL: NCT04512859
Title: Effect of Stellate Ganglion Block on Cerebral Vasospasm in Patients With Emergency Aneurysmal Subarachnoid Hemorrhage
Brief Title: Stellate Ganglion Block in Preventing Cerebral Vasospasm Secondary to Subarachnoid Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Vice Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20200630
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal; Cerebral Vasospasm
Keywords: Stellate Ganglion Block; Subarachnoid Hemorrhage; Cerebral Vasospasm; Transcranial Doppler Ultrasonography
MeSH Terms: conditions — Subarachnoid Hemorrhage; Vasospasm, Intracranial

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stellate Ganglion Block (Experimental): Experimental patients will receive a stellate ganglion block with 0.25% ropivacaine 10mL on the same side of vasospasm at the level of the sixth cervical vertebrae (C6) before surgery.
  Patients were then assessed using transcranial Doppler
  Interventions: Procedure: Stellate Ganglion Block
- No Stellate Ganglion Block (Placebo Comparator): patients will receive a stellate ganglion block with 0.9% saline 10mL on the same side of vasospasm at the level of the sixth cervical vertebrae (C6) before surgery.
  Patients were then assessed using transcranial Doppler
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Stellate Ganglion Block — Stellate ganglion block under ultra-guide will be administered using 0.25% ropivacaine 10mL
  Arms: Stellate Ganglion Block
Procedure: Placebo — Stellate ganglion block under ultra-guide will be administered using 0.9% saline 10mL
  Arms: No Stellate Ganglion Block

SUMMARY:
To investigate whether the stellate ganglion block is helpful in relieving cerebral vasospasm during aneurysmal coil embolism surgery. The effect was assessed by Transcranial Doppler (TCD).

ELIGIBILITY:
Inclusion Criteria:

* 1.Emergency patients with subarachnoid hemorrhage caused by ruptured aneurysm, aged 18-65 years; 2. ASA : II-IV grade, Hunt-Hess : I-III grade 3. For the first case, the operation time is within 24 hours. 4.After signing informed consent, underwent interventional intravascular embolization

Exclusion Criteria:

* 1. Patients with severe bleeding disorders; 2. Patients with trauma and local infection risk in the nerve block area; 3. Patients with previous aneurysm surgery and unruptured aneurysm; 4. Aneurysm located in middle cerebral artery; 5. Patients with unconsciousness cannot cooperate with the block operation; 6. Those with a history of mental illness and epilepsy; 7. Those who have a history of severe cardiovascular and cerebrovascular diseases and severe organ diseases;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of cerebral vasospasm | Change from baseline at 5day,after subarachnoid hemorrhage